CLINICAL TRIAL: NCT05733169
Title: Pre-calculation for Frequency Lowering With Hearing Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5937
Record Dates: First submitted 2023-01-27; First posted 2023-02-17 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Frequency Lowering

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hearing impaired group (Experimental): The hearing impaired group will compare the reference condition with the intervention condition.
  Interventions: Other: Frequency lowering intervention; Other: Frequency lowering reference

INTERVENTIONS:
Other: Frequency lowering intervention — Modified parametrization of the current frequency lowering parametrization.
  Other Names: Intervention condition
Other: Frequency lowering reference — Current frequency lowering parametrization
  Other Names: Reference condition

SUMMARY:
Perceptual evaluation of the parametrization and pre-calculation of frequency lowering requires the participation of subjects with hearing loss.

ELIGIBILITY:
Inclusion Criteria:

* Experienced hearing aid user (minimum use duration 1 year)
* Adult (minimum age: 18 years),
* Experience with frequency lowering,
* Hearing thresholds with N5-N7, S1, S2, S3 hearing loss
* Symmetrical hearing loss (difference between ears <= 10 dB for 1kHz-6kHz) ,
* Sensorineural hearing loss,
* Air Conduction - bone conduction gap <= 10 dB,
* Written and spoken German,
* Ability to understand instruction,
* Ability to describe listening experiences,
* Ability to attend to the appointments,
* Ability to fill in a questionnaire conscientiously
* Healthy outer ear (without previous surgical procedures)
* Hearing loss within the fitting ranges of the investigational product,
* Informed consent as documented by signature.

Exclusion Criteria:

* Clinical contraindications deformity of the ear (closed ear canal
* or absence of pinna),
* Not willing to wear the hearing aid,
* Fluctuating hearing that could influence the results,
* Contraindications to the MD in this study, e.g. known hypersen-sitivity or allergy to the investigational product,
* Limited mobility and not in the position to attend all appoint-ments,
* Limited ability to describe listening impressions/experiences and the use of the hearing aid,
* Inability to produce a reliable hearing test result,
* Massively limited dexterity,
* Known psychological problems,
* Known central hearing disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Measurement of sound quality and audibility of high-frequency sounds for hearing-impaired subjects with the new parametrization compared to the current implementation of the parametrization. | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Sonova AG, Stäfa, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No